CLINICAL TRIAL: NCT03071783
Title: Intra-operative Feed Back on Traction Force During Vacuum Extraction: a Randomized Control Study of Mid and Low Metal Cup Deliveries.
Brief Title: Intra-operative Feed Back on Traction Force During Vacuum Extraction: Safe Vacuum Extraction Alliance
Acronym: SVEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Magnus Westgren, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KI-Clintec-SVEA
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Hypoxic Ischemic Encephalopathy; Neonatal Convulsions; Subgaleal Hematoma
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vacuum extraction intelligent system (Experimental): Measurement and intra-operative feed back of vacuum extraction data: notification signal based an algorithm calculation using traction force (peak and time force integral) and time.
  Interventions: Device: Vacuum extraction intelligent system
- conventional (No Intervention): conventional handle

INTERVENTIONS:
Device: Vacuum extraction intelligent system — Vacuum extraction intelligent system - this is the intervention
  Arms: Vacuum extraction intelligent system

SUMMARY:
The objective of the clinical investigation is to test whether intra-operative traction force feed back during vacuum extraction leads to a significant decrease in incidence of brain damage in neonates.

By randomization, half of the vacuum extraction patients will be assigned to delivery using a new intelligent handle for vacuum extractions, and half will be assigned to conventional method without traction force measurement.

DETAILED DESCRIPTION:
The most common indications for vacuum extraction are dystocia and/or fetal asphyxia. The safety of assisted vaginal delivery with vacuum extraction has been discussed since its introduction almost fifty years ago. Serious complications such as asphyxia, intracranial hemorrhage and seizures are overrepresented at vacuum extraction compared to spontaneous vaginal delivery.

Little has been done to improve the procedure since the introduction. Safety measures recommended include restricting total time and number of pulls, a full 34 week gestation, and station of the head at the spines or below. A general advice is also to avoid excessive traction force. There is no general agreement to what a safe traction force might be. With exceeding force there seems to be an increased risk for rupture of the sagittal sinus and tearing of the falx at its attachment to the tentorium. Furthermore, when the fetal head is becoming exceedingly elongated and flattened, and as the cup pops off it might cause damage to the brain and blood vessels.

During the procedure the obstetrician is under significant stress and the subjective element of the evaluation of traction force is a concern. The difficult decision of whether to continue a heavy extraction or abort the operation is made under stressful conditions and based mostly on subjective impressions.

To provide the obstetrician with more objective information, the investigators developed a new device consisting of an intelligent handle hooked to the chain of a regular metal cup.

ELIGIBILITY:
Inclusion Criteria:

* Medical or social reasons for vacuum extraction with a metal cup, gestational age ≥37+0 weeks, singleton, cephalic

Exclusion Criteria:

* Multiple pregnancy, breech presentation, gestational age <37+0

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2016-04-01; Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Composite neonatal brain damage | From start of extraction through 28 days after delivery (or until discharge from the hospital)
  Composite consists of: Hypoxic ischemic encephalopathy (HIE), intracranial hemorrhage (ICH), seizures, perinatal mortality and subgaleal hematoma as routinely diagnosed in patient chart

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Westgren, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] MALMSTROM T. The vacuum extractor, an obstetrical instrument. I. Acta Obstet Gynecol Scand Suppl. 1957;36(suppl 3):5-50. No abstract available. PMID 13497632
- [Background] Moolgaoker AS, Ahamed SO, Payne PR. A comparison of different methods of instrumental delivery based on electronic measurements of compression and traction. Obstet Gynecol. 1979 Sep;54(3):299-309. PMID 471369
- [Background] Towner DR, Ciotti MC. Operative vaginal delivery: a cause of birth injury or is it? Clin Obstet Gynecol. 2007 Sep;50(3):563-81. doi: 10.1097/GRF.0b013e31811eaa39. PMID 17762410
- [Background] Whitby EH, Griffiths PD, Rutter S, Smith MF, Sprigg A, Ohadike P, Davies NP, Rigby AS, Paley MN. Frequency and natural history of subdural haemorrhages in babies and relation to obstetric factors. Lancet. 2004 Mar 13;363(9412):846-51. doi: 10.1016/S0140-6736(04)15730-9. PMID 15031028
- [Result] Pettersson K, Ajne J, Yousaf K, Sturm D, Westgren M, Ajne G. Traction force during vacuum extraction: a prospective observational study. BJOG. 2015 Dec;122(13):1809-16. doi: 10.1111/1471-0528.13222. Epub 2015 Jan 5. PMID 25558833
- [Derived] Romero S, Pettersson K, Yousaf K, Westgren M, Ajne G. Perinatal outcome after vacuum assisted delivery with digital feedback on traction force; a randomised controlled study. BMC Pregnancy Childbirth. 2021 Feb 26;21(1):165. doi: 10.1186/s12884-021-03604-z. PMID 33637058